CLINICAL TRIAL: NCT03564574
Title: To Study the Effects of Lipid Emulsion on Hemodynamics in Organophosphate Compound Poisoning
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, Bharath A. Chhabria, Doctor, Post Graduate Institute of Medical Education and Research, Chandigarh
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: bharath_thesis
Record Dates: First submitted 2016-05-03; First posted 2018-06-21 (Actual); Last update posted 2018-06-21 (Actual); Status verified 2018-06

CONDITIONS: Organophosphate Poisoning
MeSH Terms: conditions — Organophosphate Poisoning | interventions — Fat Emulsions, Intravenous

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Study group (Experimental): Inclusion criteria
  1. History of consumption of OP compound.
  2. Symptom complex consistent with OP poisoning
  3. Age > 18 years
  4. Informed consent from the patient or next kin.
  Exclusion criteria
  1. History of combined poisoning with a non OP compound.
  2. All other patients not fitting in the organophosphate symptom complex.
  3. Patients with underlying liver and kidney disease.
  4. History suggestive of acute pancreatitis in the past.
  All patients with history and clinical features of OP compound poisoning admitted to the emergency department in PGIMER during the study period, meeting the inclusion, exclusion criteria and who gave consent were enrolled in the study.
  Intervention : Administration of 100mL of 20% Lipid emulsion to all patients in the study group
  Interventions: Combination Product: Lipid Emulsion
- Historic controls (No Intervention): The control arm The study group was compared with data of patients admitted for OP poisoning between the years 2013 and 2014 ( 2 calendar years), fulfilling the inclusion and exclusion criteria as stated above.

INTERVENTIONS:
Combination Product: Lipid Emulsion — All patients in the 'Study group' received a single dose of 100 ml of 20 percent Lipid emulsion as an infusion over 1 hour along with routine treatment as per institution protocols. Atropine was administered to patients by doubling dose method, which comprised of administering atropine starting from 2mg and to double the dose and administer till complete atropinization. Following this an infusion of 10 percent of the atropinizing dose was given every hour. Patients were evaluated using a standardized clinical interview, physical examination, laboratory tests.
  Other Names: Intralipid 20 percent
  Arms: Study group

SUMMARY:
To Study the Effects of Lipid Emulsion on Hemodynamics in Organophosphate Compound Poisoning Objectives: To study the effect of administration of intravenous lipid emulsion on hemodynamic parameters, incidence of adverse effects in patients with organophosphate poisoning.

Background: Lipid emulsion has been used to revert toxicities of lipophilic drugs, toxins (especially lignocaine) and in critically ill patients. Though the safety has been established, the effect on hemodynamics in Organophosphate (OP) poisoned patients has never been studied. Hence this study is underway to fill those lacunae and evaluate the safety profile of lipid emulsion in organophosphate poisoned patients.

Methodology: The study is a prospective open label pilot study, which is underway at a tertiary care hospital in North India. Patients with history and clinical features of OP poisoning meeting the inclusion and exclusion parameters are being treated according to institutional protocols. Along with routine treatment a single dose of 20% lipid emulsion is being administered on admission to patients after obtaining consent. Patients are being followed up till discharge or death. Hemodynamic parameters and adverse effects following lipid emulsion administration are being studied over various intervals of time.

DETAILED DESCRIPTION:
Methods A prospective open label pilot study was conducted with an aim to study the safety and effects of 20% lipid emulsion in OP compound poisoning. The objectives were to study the effects on hemodynamic parameters, the effect on morbidity, mortality and the occurrence of adverse events.

All patients, ≥ 13 years, with history of consumption of OP compound and clinical features of mild, moderate or severe OP compound poisoning as per the Peradeniya score (Table 1), admitted to the emergency department during the study period from September 2015 - December 2016 were included after written informed consent. Consent was obtained from the nearest kin if the presentation was with altered mental state. The recruitment began after approval from the institute's ethics committee.

Patients with chronic liver or kidney disease, history of acute or chronic pancreatitis in the past, those with combined poisoning with non OP compounds and asymptomatic patients were not included.

At presentation, detailed history was sought and subjects were examined for signs and symptoms of OP poisoning. Vital parameters (pulse rate, blood pressure, and respiratory rate) were noted. Blood samples were drawn for assessing baseline electrolytes, renal functions, haematological parameters and serum amylase. All patients received a single dose of 100mL of 20% lipid emulsion as an intra-venous infusion over 1 hour along with routine treatment as per institution protocols. Atropine was administered to patients by doubling dose method, which comprised of administering atropine starting from 2mg and to double the dose and administer till complete atropinization. Following this an infusion of 10-20 percent of the atropinizing dose was given every hour. In view of the controversial role of pralidoxime, it was not included in the study. The cases were followed up until recovery/death.

The patients were under observation for their vital signs, pupil size, fasciculation, respiratory crackles, amount of oral secretions and, if intubated, tracheal secretion. In addition they underwent monitoring of vital parameters every ten minutes during the course of lipid administration for the first thirty minutes followed by every fifteen minutes during the next 2 hours and every 2nd hourly thereafter.

Hemodynamic parameters, haematological, biochemical parameters, adverse effects and outcomes were compared at various intervals of time following administration of lipid emulsion, up to 72 hours, with those at the baseline; hemodynamic parameters were also compared with historic controls.

The primary outcome was to study the change in hemodynamic parameters (pulse rate, systolic blood pressure, mean arterial pressure and respiratory rate) after delivery of lipid emulsion in OP poisoned individuals up to 72 hours and compare any changes in the hemodynamic parameters with that of historic controls.

Secondary outcomes were to study the effects on case fatality (in-hospital until discharge or death), morbidity (duration of hospitalization, duration of mechanical ventilation, dose of atropine given) and the occurrence of complications including those related to lipid emulsion and hospital acquired infections.

ELIGIBILITY:
Inclusion criteria

1. History of consumption of OP compound.
2. Symptom complex consistent with OP poisoning
3. Age > 18 years
4. Informed consent from the patient or next kin.

Exclusion criteria

1. History of combined poisoning with a non OP compound.
2. All other patients not fitting in the organophosphate symptom complex.
3. Patients with underlying liver and kidney disease.
4. History suggestive of acute pancreatitis in the past.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Significant change in pulse from baseline to 72 hours after admission | Date of admission up to 72 hours
  The primary outcome was to study the change in
  1.Pulse (beats/min) after delivery of lipid emulsion in OP poisoned individuals at various intervals of time from time of admission to 72 hours after administration of lipid emulsion and compare the same data with historic controls
Significant change in systolic blood pressure from baseline to 72 hours after admission | Date of admission up to 72 hours
  The primary outcome was to study the change in 2.Systolic blood pressure (mm Hg) after delivery of lipid emulsion in OP poisoned individuals at various intervals of time from time of admission to 72 hours after administration of lipid emulsion and compare the same data with historic controls
Significant change in oxygen arterial saturation from baseline to 72 hours after admission | Date of admission up to 72 hours
  Change in arterial oxygen saturation (SpO2) in percentage
Adverse effects | Date of admission until discharge/death of subjects up to 1 month
  Incidence of adverse reactions in percentage
Significant change in diastolic blood pressure from baseline to 72 hours after admission | Date of admission up to 72 hours
  The primary outcome was to study the change in 5. Diastolic blood pressure (mm Hg) after delivery of lipid emulsion in OP poisoned individuals at various intervals of time from time of admission to 72 hours after administration of lipid emulsion and compare the same data with historic controls
Significant change in mean arterial pressure from baseline to 72 hours after admission | Date of admission up to 72 hours
  The primary outcome was to study the change in 6. Mean arterial pressure (mm Hg) after delivery of lipid emulsion in OP poisoned individuals at various intervals of time from time of admission to 72 hours after administration of lipid emulsion and compare the same data with historic controls

SECONDARY OUTCOMES:
Effect on case fatality and morbidity | Admission to the hospital till time of discharge up to 1 month
  Secondary outcomes were to study the effects on
  1. All cause mortality (in-hospital until discharge or death), that is the case fatality and morbidity in terms of duration of hospitalization in days, duration of mechanical ventilation in days, dose of atropine given in milligram an The data was compared with historic controls

CONTACTS AND LOCATIONS:
Locations (1):
- Pgimer, Chandigarh, India

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Chhabria BA, Bhalla A, Shafiq N, Kumar S, Dhibar DP, Sharma N. Lipid emulsion for acute organophosphate insecticide poisoning - a pilot observational safety study. Clin Toxicol (Phila). 2019 May;57(5):318-324. doi: 10.1080/15563650.2018.1520997. Epub 2018 Oct 11. PMID 30307350